CLINICAL TRIAL: NCT00471458
Title: Follow-up Study of Hyperthyroid Patients Treated With RAI in 1965-2002: Morbidity in Long-Term Follow-up
Brief Title: Follow-up Study of the RAI-Treated Hyperthyroid Patients
Status: Completed | Type: Observational
Sponsor: Tampere University (Other)
Other Study IDs: R02134
Record Dates: First submitted 2007-05-09; First posted 2007-05-10 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Hyperthyroidism; Cardiovascular Diseases; Atrial Fibrillation
Keywords: Radioiodine; Hyperthyroidism; Morbidity; Cardiovascular diseases
MeSH Terms: conditions — Hyperthyroidism; Cardiovascular Diseases; Atrial Fibrillation

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Previous studies of hyperthyroid patients suggest that they remain at increased risk of cardiovascular morbidity after restoring euthyroidism.

The study objective is to compare the rate and causes of hospitalization of hyperthyroid patients treated with radioactive iodine (RAI) with those of an age- and gender-matched reference population in a long-term follow-up study.

DETAILED DESCRIPTION:
A population-based cohort study was conducted among 2611 hyperthyroid patients treated with RAI between 1969 and 2002 in Tampere University Hospital, and among 2611 reference subjects. A reference group was randomly selected, with an age- and gender-matched control subject identified for each patient from the Population Register Centre. The control subject had to be alive at the time when the patient received the first RAI treatment.

The causes of hospitalization as well as the diagnosis and date of hospital admission were obtained from the nationwide Hospital Discharge Register (HILMO) maintained by the Research and Development Centre for Welfare and Health (STAKES) using a computerized record linkage, with the personal identification number as the key. The HILMO database covers all dates and causes of hospitalization (hospital admission requiring an overnight stay) of the Finnish citizens since January 1969. New events were analyzed as the main outcome, including only the first hospitalization due to a given indication. The special focus was on the cardiovascular morbidity.

ELIGIBILITY:
Inclusion Criteria:

* Patients: Radioiodine treatment for hyperthyroidism given in the Tampere University Hospital between January 1969 and June 2002
* Controls: age- and gender-matched control subject identified for each patient from the Population Register Centre. The control subject had to be alive at the time when the patient received the first RAI treatment

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 5222 (Actual)
Dates: Start 1969-01; Study Completion 2003-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Saara Metso, MD, Principal Investigator — Tampere University Hospital, Department of Internal Medicine, FIN-33521 Tampere, Finland; Pia Jaatinen, MD, PhD, Study Director — Medical School, University of Tampere, Tampere, FINLAND; Jorma Salmi, MD, PhD, Study Director — Tampere University Hopsital, Department of Internal Medicine, FIN-33521 TAMPERE, FINLAND
Locations (1):
- Tampere University Hospital, Department of Internal Medicine, Tampere, Finland

REFERENCES:
- [Background] Metso S, Jaatinen P, Huhtala H, Luukkaala T, Oksala H, Salmi J. Long-term follow-up study of radioiodine treatment of hyperthyroidism. Clin Endocrinol (Oxf). 2004 Nov;61(5):641-8. doi: 10.1111/j.1365-2265.2004.02152.x. PMID 15521969
- [Background] Metso S, Auvinen A, Huhtala H, Salmi J, Oksala H, Jaatinen P. Increased cancer incidence after radioiodine treatment for hyperthyroidism. Cancer. 2007 May 15;109(10):1972-9. doi: 10.1002/cncr.22635. PMID 17393376
- [Background] Metso S, Jaatinen P, Huhtala H, Auvinen A, Oksala H, Salmi J. Increased cardiovascular and cancer mortality after radioiodine treatment for hyperthyroidism. J Clin Endocrinol Metab. 2007 Jun;92(6):2190-6. doi: 10.1210/jc.2006-2321. Epub 2007 Mar 20. PMID 17374710